CLINICAL TRIAL: NCT05897866
Title: Sayed Issa's Hybrid Limited Shoulder Surgical Management (HLSSM)
Brief Title: Sayed Issa's Hybrid Shoulder Arthroscopic-Open Surgical Management (HSSM)
Acronym: HLSSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Issa, Abdulhamid Sayed, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sayed Issa's HLSSM; HLSSM (Other: Dr. Abdulhamid Sayed Issa Clinic)
Record Dates: First submitted 2023-05-12; First posted 2023-06-09 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2020-09

CONDITIONS: Shoulder Impingement Syndrome; Adhesive Capsulitis; Rotator Cuff Tear; Hill-Sachs Lesion; Frozen Shoulder; Tendinopathy
Keywords: Shoulder; Shoulder approach; Lateral Shoulder approach; Shoulder impingement syndrome; Rotator cuff tendinopathy; Adhesive capsulitis; Frozen shoulder syndrome; MLSA; Shoulder arthroscopy; Mini Lateral Shoulder Approach; Second Sayed Issa's Approach; Hill-sachs lesion; mini-incision release; Tendinopathy; arthroscopy; tendon injuries
MeSH Terms: conditions — Shoulder Impingement Syndrome; Bursitis; Rotator Cuff Injuries; Bankart Lesions; Tendinopathy; Tendon Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Issa3 (Experimental): Dr.A.Sayed Issa and his team
  Interventions: Procedure: Sayed Issa's Hybrid Shoulder Arthroscopic-Open Surgical Management

INTERVENTIONS:
Procedure: Sayed Issa's Hybrid Shoulder Arthroscopic-Open Surgical Management — Using Arthroscopy and then Limited Opening by Mini Lateral Shoulder Approach (MLSA) for the shoulder surgery.
  Other Names: Sayed Issa's HSSM

SUMMARY:
Sayed Issa's Hybrid Shoulder Arthroscopic-Open Surgical Management (HSSM) is a limited lateral approach to the shoulder arthroscopically guided. Which achieves less surgical trauma and smaller surgical incision than even in Mini Lateral Shoulder Approach (MLSA).

DETAILED DESCRIPTION:
After making a full clinical, X-rays and MRI examinations of the shoulder, and finding Shoulder Impingement Syndrome, Adhesive Capsulitis, Rotator Cuff Tear, or Hill-Sachs lesion, we decide to manage the problem surgically We can survey the shoulder from the inside and determine the shape, size and the exact position of the defect by shoulder arthroscopy.

The patient is operated on under general anesthesia; shoulder arthroscopy can be performed in the lateral decubitus or beach chair position which is the basic shoulder arthroscopy (Beach Chair Patient Positioning).

After identifying the full characteristics of the lesion, we go for Mini Lateral Shoulder Approach (MLSA), as known as Second Sayed Issa's Approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with Shoulder Impingement Syndrome refractory to conservative treatment and local steroid injection
* Patients presented with Adhesive Capsulitis and Frozen Shoulder Syndrome refractory to conservative treatment and local steroid injection
* Patients without femur head immigration on X-ray
* Patients with injury for one month to six months maximum

Exclusion Criteria:

* Patients with femur head immigration on X-ray
* Patients with injury for more than six months
* Uncontrolled diabetes mellitus type 1 and 2
* Patients with non controlled Vascular hypertension
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Less open surgery trauma | 25 minutes to 45 minutes,
  Directly going to the goal lesion with less expansion

SECONDARY OUTCOMES:
Smaller surgical incision than MLSA | Less than 5 cm
  Directly going to the goal lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdulhamid Sayed Issa Clinic, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: Yes
URL: http://www.asayedissa.com

REFERENCES:
- See also: Related Info — http://asayedissa.com